CLINICAL TRIAL: NCT01323855
Title: A Study to Assess Pharmacokinetics of Preladenant in Subjects With Chronic Renal Impairment
Brief Title: A Study to Assess Pharmacokinetics (PK) of Preladenant in Participants With Chronic Renal Impairment (CRI) (P06512)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06512; 2010-023063-18 (EudraCT Number); MK-3814-031 (Other: Merck)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: Severe Renal Impairment (Experimental): Participants with severe CRI, defined as creatinine clearance of <30 mL/min/1.73 m^2, were treated with a single tablet of 5 mg preladenant, administered orally
  Interventions: Drug: Preladenant
- Part 2: Moderate Renal Impairment (Experimental): Participants with moderate CRI defined as creatinine clearance of ≥30 and <50 mL/min/1.73 m^2, were treated with a single tablet of 5 mg preladenant, administered orally
  Interventions: Drug: Preladenant
- Part 2: Mild Renal Impairment (Experimental): Participants with mild CRI, defined as creatinine clearance of ≥50 and ≤80 mL/min/1.73m^2, were treated with a single tablet of 5 mg preladenant, administered orally
  Interventions: Drug: Preladenant
- Part 1: Normal Renal Function (Experimental): Participants with normal renal function, defined as creatinine clearance of >80 mL/min/1.73 m^2, were treated with a single tablet of 5 mg preladenant, administered orally
  Interventions: Drug: Preladenant
- Part 2: Normal Renal Function (Experimental): Participants with normal renal function, defined as creatinine clearance of >80 mL/min/1.73 m^2, were treated with a single tablet of 5 mg preladenant, administered orally
  Interventions: Drug: Preladenant

INTERVENTIONS:
Drug: Preladenant — After an overnight fast, a single 5 mg dose, (1 x 5 mg tablet) was administered orally
  Other Names: SCH 420814

SUMMARY:
This is a two part study to compare the PK of preladenant administered to participants with CRI to the PK of preladenant administered to healthy participants. Part 1 will compare the PK of participants with severe CRI to healthy participants. Part 2 will compare the PK of participants with moderate CRI and participants with mild CRI to healthy participants. The primary hypotheses are that the plasma area under the concentration-time curve from time 0 to infinity after single dosing (AUC0-∞) of preladenant in participants with either severe, moderate or mild CRI is similar to that of matched healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) between 19 to 34 kg/m^2, inclusive
* Has mild to severe CRI and not on dialysis (Participants with normal renal function are to be matched to subjects with renal impairment)
* Clinical laboratory tests, electrocardiogram, and vital signs within normal ranges
* Free of any clinically significant disease that would interfere with the study evaluations (except related to his/her renal disease and comorbid conditions)

Exclusion Criteria:

* Females who are pregnant, intend to become pregnant (within 3 months of ending the study), or are nursing/breastfeeding
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* Had a renal transplant or are on dialysis
* Has a history of any infectious disease within 4 weeks
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has donated blood or had a blood transfusions in the past 60 days
* Has demonstrated allergic reactions (eg, food, drug, atopic reactions or asthmatic episodes) which could interfere with their ability to participate in the trial
* Has a history of malignancy
* Has evidence of suicidality or is at risk for self-harm or harm to others

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-03-28 (Actual); Primary Completion 2011-11-29 (Actual); Study Completion 2011-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female adults with different degrees of renal impairment along with matched healthy adults with normal renal function were selected for this study.
Groups:
- Part 1: Severe Renal Impairment: Participants with severe chronic renal impairment (CRI), defined as creatinine clearance of <30 mL/min/1.73 m^2, were treated with a single tablet of 5 mg preladenant, administered orally
Period: Overall Study
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function
Started | 9 | 9 | 8 | 9 | 11
Completed | 9 | 9 | 8 | 9 | 11
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function | Total
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (12.4) | 66.9 (7.8) | 63.3 (7.6) | 59.3 (11.3) | 67.4 (4.0) | 63.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 3 | 5 | 20
  Male | 6 | 5 | 3 | 6 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) After Single Dosing With Preladenant for Participants With Severe CRI Versus Healthy Matched Controls
Description: Blood samples were taken at the following timepoints: pre-dose, 0.25, 0.50, 0.75, 1, 2, 4, 6, 12, 16, 24, 30, 36 and 48 hours postdose in order to determine the AUC0-∞ of preladenant
Time Frame: Pre-dose to 48 hours post-dose
Population: Four participants with severe CRI, and two matched healthy participants with insufficient terminal phase data to allow adequate characterization, were not analyzed. As only participants with severe CRI are presented, participants with mild or moderate CRI or their corresponding healthy matched controls were not analyzed in this outcome measure
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function
Number analyzed (Participants) | 5 | 0 | 0 | 7 | 0
ng.hr/mL | 160.53 [81.13 to 317.62] |  |  | 135.12 [77.83 to 234.56] |
Statistical Analysis 1: Comparison: Part 1: Severe Renal Impairment vs Part 1: Normal Renal Function; Test type: Non-Inferiority or Equivalence — Geometric Mean Ratio (GMR) is contained within the interval [0.50, 2.00]; GMR = 1.19, 90% CI 2-sided [0.54 to 2.62] — Severe CRI/Healthy

2. Primary Outcome: AUC0-∞ After Single Dosing With Preladenant for Participants With Moderate CRI Versus Healthy Matched Controls
Description: as for outcome 1
Time Frame: Pre-dose to 48 hours post-dose
Population: One participant with moderate CRI, and two matched healthy participants with insufficient terminal phase data to allow adequate characterization, were not analyzed. As only participants with moderate CRI are presented, participants with mild or severe CRI or their corresponding healthy matched controls were not analyzed in this outcome measure
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function
Number analyzed (Participants) | 0 | 8 | 0 | 0 | 5
ng.hr/mL |  | 197.43 [99.12 to 393.25] |  |  | 152.18 [67.65 to 342.34]
Statistical Analysis 1: Comparison: Part 2: Moderate Renal Impairment vs Part 2: Normal Renal Function; Test type: Non-Inferiority or Equivalence — GMR is contained within the interval [0.50, 2.00]; GMR = 1.30, 90% CI 2-sided [0.59 to 2.87] — Moderate CRI/Healthy

3. Primary Outcome: AUC0-∞ After Single Dosing With Preladenant for Participants With Mild CRI Versus Healthy Matched Controls
Description: as for outcome 1
Time Frame: Pre-dose to 48 hours post-dose
Population: One participant with mild CRI, and two matched healthy participants with insufficient terminal phase data to allow adequate characterization, were not analyzed. As only participants with mild CRI are presented, participants with severe or moderate CRI or their corresponding healthy matched controls were not analyzed in this outcome measure
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function
Number analyzed (Participants) | 0 | 0 | 7 | 0 | 4
ng.hr/mL |  |  | 275.50 [183.51 to 413.61] |  | 104.66 [65.54 to 167.15]
Statistical Analysis 1: Comparison: Part 2: Mild Renal Impairment vs Part 2: Normal Renal Function; Test type: Non-Inferiority or Equivalence — GMR is contained within the interval [0.50, 2.00]; GMR = 2.63, 90% CI 2-sided [1.38 to 5.04] — Mild CRI/Healthy

ADVERSE EVENTS:
Time Frame: Up to Day 7
Description: All enrolled participants
Arm/Group | Part 1: Severe Renal Impairment | Part 2: Moderate Renal Impairment | Part 2: Mild Renal Impairment | Part 1: Normal Renal Function | Part 2: Normal Renal Function
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 1/8 | 0/9 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Severe Renal Impairment (N=9) | Part 2: Moderate Renal Impairment (N=9) | Part 2: Mild Renal Impairment (N=8) | Part 1: Normal Renal Function (N=9) | Part 2: Normal Renal Function (N=11)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.